CLINICAL TRIAL: NCT05875350
Title: Efficacy of Low Dose Intraligamental Local Anesthesia as an Alternative for Infiltration Technique for Extraction of Grade II Mobility Maxillary Molars: Double Blind Randomized Clinical Trial
Brief Title: Intraligamental Local Anesthesia Versus Infiltration Technique for Extraction of Grade II Mobility Maxillary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Tarek Abdelbarry, Lecturer of Oral and Maxillofacial Surgery, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 716
Record Dates: First submitted 2023-05-12; First posted 2023-05-25 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraligamental local anesthetic injection (Experimental)
  Interventions: Procedure: Intraligamental local anesthetic injection
- Buccal infiltration local anesthetic injection (No Intervention)

INTERVENTIONS:
Procedure: Intraligamental local anesthetic injection — The intraligamental technique was administered using ligajet intraligamentary jet injector (Micro Mega Company) containing Articaine hydrochloride 4% with adrenaline 1:200000 (ArtPharma Dent, inc, Egypt)
  Arms: Intraligamental local anesthetic injection

SUMMARY:
The study aims to assess the use of intraligamental local anesthetic injection compared to buccal infiltration for extraction of maxillary molars suffering grade II mobility in terms of pain control and extraction duration.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients (class I category according to American society of anesthesiologists )
* Age range: 20 - 60 years of age,
* Either genders who are seeking dental extraction of maxillary molar teeth diagnosed with grade II mobility.

Exclusion Criteria:

* Patients with tooth that require trans osseous extraction
* Badly broken down coronal structure of the tooth to be extracted
* Patients with significant medical conditions
* Alcoh intake
* Patients on drugs that affect the central nervous systems
* Patients who reported the use of drugs that might interfere with pain sensitivity
* Pregnant or lactating women
* Patients who suffer from hypersensitivity to local anesthetics or non-steroidal anti-inflammatory drugs (NSAIDs).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Pain using visual analogue scale | immediately after injection
  visual analogue scale (VAS) was used in which a pain score was recorded for each patient just after local anesthetic adminstration. The VAS score ranges from 0 (no pain) to 10 (extreme unbearable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided